CLINICAL TRIAL: NCT01412606
Title: Endometrial Scratching in Couples With Unexplained Subfertility
Acronym: ESUS
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Ahmed Gibreel, Dr, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AG2
Record Dates: First submitted 2011-08-08; First posted 2011-08-09 (Estimated); Last update posted 2012-08-30 (Estimated); Status verified 2012-08

CONDITIONS: Subfertility
Keywords: Unexplained infertility-endometrial scratching; effect of endometrial biopsy (scratching) on clinical pregnancy rates in women with unexplained infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Scrathcing (Experimental): scratching of endometrium on day 21-26 of a spontaneous menstrual cycle
  Interventions: Procedure: scratching
- Control (Placebo Comparator): Uterine sounding on day 21-26 of a spontaneous menstrual cycle
  Interventions: Procedure: scratching

INTERVENTIONS:
Procedure: scratching — scratching endometrium on day 21-26 of a spontaneous menstrual cycle

SUMMARY:
Endometrial scratching in luteal phase of a spontaneous menstrual cycle may increase pregnancy rate in women with unexplained infertility.

ELIGIBILITY:
Inclusion Criteria:

* women aged between 20 and 39 years with at least one year of infertility
* regular menstruation with the length of the cycle between 22-34 days and ovulation confirmed by appropriately timed mid-luteal progesterone
* fertile semen variables
* bilateral tubal patency (demonstrated by laparoscopy or hysterosalpingography).

Ages: 20 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 105 (Actual)
Dates: Start 2009-07; Primary Completion 2010-12 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Clinical pregnancy rate | 6 months

SECONDARY OUTCOMES:
miscarriage rate | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Gibreel, MD, Principal Investigator — Mansoura University
Locations (1):
- Mansoura University Teaching Hospital Gynecology outpatient clinic, Al Mansurah, Egypt

REFERENCES:
- [Derived] Gibreel A, Badawy A, El-Refai W, El-Adawi N. Endometrial scratching to improve pregnancy rate in couples with unexplained subfertility: a randomized controlled trial. J Obstet Gynaecol Res. 2013 Mar;39(3):680-4. doi: 10.1111/j.1447-0756.2012.02016.x. Epub 2012 Oct 29. PMID 23106834